CLINICAL TRIAL: NCT07318168
Title: Randomized Controlled Pilot Trial of a Brief Psycho-educational Intervention to Enhance Maternal Reflective Functioning in the Early Postpartum Among First-Time Mothers
Brief Title: Brief Psycho-educational Intervention to Enhance Maternal Reflective Functioning in the Early Postpartum Among Primiparous: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Lee Barel Refaeli, Lecturer and PhD candidate, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UHaifa-pilot-womenpostnatal-LB
Record Dates: First submitted 2025-12-02; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Period; Maternal Mental Health; Parenting / Maternal Behavior; Primiparity (First-Time Mothers); Depressive Symptoms, Postpartum
Keywords: Maternal Reflective Functioning (RF); Mentalization / Parental Mentalization; First-Time Mothers / Primiparous; Early Postpartum; Psychoeducational Group Intervention; Telehealth / Zoom; FMSS-RF; PRFQ; EPDS; Emotion Regulation (ERQ); Feasibility / Acceptability; Israel / University of Haifa
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 two-arm parallel trial comparing a brief psycho-educational group intervention versus wait-list control among first-time mothers. Assessments at baseline (T1) and post-intervention (T2 ~4-5 weeks after T1). Outcome assessors (FMSS-RF coders) were blinded to group and time.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors (FMSS-RF coders) were blinded to group assignment and time point; participant blinding was not feasible for a behavioral program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Four weekly 90-minute online psycho-educational group sessions targeting maternal reflective functioning (RF), with brief home practice; make-up allowed for one missed session.
  Interventions: Behavioral: Thinking Emotions - Postpartum RF Group
- Wait-List Control (No Intervention): Participants received usual care and were offered the same group program after completion of the post-intervention assessment (T2).

INTERVENTIONS:
Behavioral: Thinking Emotions - Postpartum RF Group — Brief psycho-educational program to enhance maternal reflective functioning (RF): four weekly 90-minute Zoom group sessions led by a trained clinician; components include recognizing mental states, perspective-taking, reading infant cues, emotion-regulation strategies, and repair of mismatches; brief home practices between sessions.
  Arms: Intervention

SUMMARY:
This randomized pilot trial tests a brief psycho-educational group program designed to enhance maternal reflective functioning (RF)-the capacity to understand one's own and the baby's behavior in terms of thoughts and feelings-among first-time mothers in the early postpartum. Primiparous women aged ≥18 years, 1-5 months postpartum, were randomized 1:1 to the intervention or a wait-list control. The intervention consists of four weekly 90-minute Zoom sessions with short home practices.

The primary outcome is interview-based RF assessed with the FMSS-RF (blind-coded) at post-intervention. Exploratory outcomes include self-reported RF (PRFQ-CMS), depressive symptoms (EPDS), emotion-regulation (ERQ-Suppression), and feasibility/acceptability indices (recruitment, retention, attendance, satisfaction).

This single-site study is conducted at the University of Haifa (Faculty of Education). If effective, the low-intensity, telehealth format may offer a scalable postpartum support option for first-time mothers.

DETAILED DESCRIPTION:
Background and Rationale. The transition to first-time motherhood is a sensitive period for women's mental health and for establishing early caregiving. Maternal reflective functioning (RF) supports sensitive caregiving and mother-infant adaptation, yet brief and scalable RF-focused postpartum supports are scarce. We developed a short psycho-educational program targeting core RF skills (identifying mental states, pausing and reflecting under stress, reading infant cues, perspective-taking, and repairing mismatches).

Objectives. (1) Evaluate feasibility and acceptability (recruitment, attendance, retention, satisfaction). (2) Estimate preliminary efficacy on maternal RF (primary) and explore effects on maternal symptoms and emotion regulation.

Design and Procedures. Community-recruited primiparous mothers (≥18 years; 1-5 months postpartum; fluent in Hebrew; internet access) completed baseline (T1) and were randomized 1:1 to Intervention versus Wait-List using a computer-generated schedule with concealed allocation. The intervention includes four weekly 90-minute Zoom sessions delivered by a trained clinician and brief home practices; make-up was offered for one missed session. Wait-list participants were offered the program after the post-intervention assessment. Masking of participants was not feasible; FMSS-RF transcripts were coded blind to group and time by trained raters (excellent inter-rater reliability). Outcomes are assessed at T1 (baseline) and post-intervention (T2; ~4-5 weeks after T1).

Measures.

Primary: Interview-based maternal RF (FMSS-RF global score) at T2.

Exploratory: PRFQ-CMS (self-report RF), EPDS (depressive symptoms), ERQ-Suppression, plus feasibility/acceptability indices.

Analysis. Pilot-level estimation emphasizes effect sizes and 95% confidence intervals. Primary analyses test the Group×Time effect on FMSS-RF (with mixed-models/ANCOVA adjusting for baseline); intention-to-treat analyses are planned alongside per-protocol sensitivity analyses.

Oversight and Transparency. Approved by the University of Haifa Ethics Committee (Faculty of Education; approval 350/21). Minimal risk; no data monitoring committee. The trial is retrospectively registered; the FMSS-RF at post-intervention is the pre-specified primary outcome, and other outcomes are labeled exploratory. De-identified materials and analysis code will be shared on OSF consistent with institutional policy.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women (first-time mothers).
* Age ≥18 years.
* 1-5 months postpartum at enrollment.
* Fluent in Hebrew and able to provide informed consent.
* Internet access and a device enabling Zoom sessions.
* Availability to attend four weekly 90-minute group sessions.

Exclusion Criteria:

* Current psychosis, bipolar manic episode, or active suicidality requiring urgent care.
* Substance dependence in the past 6 months.
* Severe cognitive/neurological condition that would preclude participation.
* Concurrent enrollment in another structured parenting/RF intervention during the trial period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in interview-based maternal reflective functioning (FMSS-RF) from baseline to post-intervention | Baseline (T1) and post-intervention at ~4-5 weeks (T2)
  FMSS transcripts are coded blind to group and time using the Reflective Functioning Scale (global RF score, 1-9, higher = better RF). Primary analysis tests the Group×Time effect (mixed models/ANCOVA adjusting for baseline); intention-to-treat alongside per-protocol.

SECONDARY OUTCOMES:
Change in self-reported parental mentalization (PRFQ-Certainty About Mental States) | Baseline (T1) and post-intervention at ~4-5 weeks (T2)
  PRFQ-CMS subscale (Likert 1-7; higher = greater certainty about mental states). Pre-specified exploratory outcome; analyzed as change from baseline and Group×Time.
Change in postpartum depressive symptoms (EPDS) | Baseline (T1) and post-intervention at ~4-5 weeks (T2)
  Edinburgh Postnatal Depression Scale (0-30; higher = more symptoms). Exploratory; analyzed as change/Group×Time.
Change in emotion-regulation - Expressive Suppression (ERQ-S) | Baseline (T1) and post-intervention at ~4-5 weeks (T2)
  ERQ Suppression subscale (Likert 1-7; higher = greater suppression). Exploratory; analyzed as change/Group×Time.
Recruitment and retention | post-intervention at ~4-5 weeks (T2)
  Recruitment rate = enrolled / eligible approached (%); Retention = % completing T2;
Attendance | Baseline+ one week post baseline, two weeks post baseline, three weeks post baseline
  Attendance = number of sessions attended (0-4)

OTHER OUTCOMES:
Number of Participants with adverse events related to participation | Baseline and 6 weeks post baseline
  Self-reported adverse events collected each session and at T2; behavioral, minimal-risk program. Count and proportion of participants reporting any AE related to participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Education, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the original consent did not include public data sharing and the dataset involves a sensitive postpartum population. Aggregate results and analysis code will be shared.

REFERENCES:
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732